CLINICAL TRIAL: NCT00563758
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study to Assess the Efficacy, Safety and Tolerability of Tegaserod 2 mg Bid vs Placebo in Patients With Chronic Constipation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW03-313 T/313; HARECCTR0500046
Record Dates: First submitted 2007-08-15; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Constipation; Chronic Disease
Keywords: Chronic constipation
MeSH Terms: conditions — Constipation; Chronic Disease | interventions — tegaserod

INTERVENTIONS:
Drug: tegaserod

SUMMARY:
Idiopathic or functional constipation is a common disorder, affecting up to 20% of the population depending on demographic factors, the sampling situation and the definitions used. Constipation is a symptom of many diseases and is a collective term, used by the patient to imply that stools are too hard, too infrequent or too difficult to pass. A recent survey conducted in Hong Kong showed a prevalence of 14% according to the Rome criteria. Based on an epidemiological study in US, there were 2.5 million annual physician visits for this problem. Exact epidemiological data however are lacking, mainly because of the difference between self-reported constipation and scientifically defined constipation.

Treatment of constipation is usually based on increased dietary fiber and supplementation with bulking agents, exercise, and habit training. However, often only partial relief is obtained, and the majority of patients use non-bulking laxatives on a regular basis without medical supervision. Chronic use of non-bulking laxatives is often inappropriate3, and may lead to side effects such as dependency and progressive tolerance, electrolyte imbalance, and, for the anthraquinones, melanosis coli. In addition, stimulant laxatives may damage the myenteric plexus4, resulting in cathartic colon5. A more appropriate approach to the therapy of constipation consists of physiologically stimulating intestinal motility.

Tegaserod, an aminoguanidine indole compound, is a representative of a new class of 5-HT4 agonists, with regard to both chemistry and pharmacology. Activation of 5-HT4 receptors triggers the release of neurotransmitters from the enteric nerves resulting in increased contractility and stimulation of the peristaltic reflex.

In animal models, tegaserod acts as a motility-enhancing agent, exerting activity throughout the gastrointestinal tract11. Tegaserod has also been shown to significantly accelerate bowel transit in healthy volunteers and in patients with constipation-predominant irritable bowel syndrome (C-IBS).

Based on the pharmacodynamic properties, tegaserod is a promotile compound suitable for the treatment associated with small and/or large bowel dysfunction e.g. constipation.

From phase III adequate and well-controlled studies in patients with C-IBS it has been shown that tegaserod was effective in relieving symptoms of C-IBS. The effect was seen as early as the first week of treatment with sustained effects over 12 weeks. Both tegaserod 4 mg/d (2 mg bid) and 12 mg/d (6 mg bid) significantly increased bowel frequency and decreased stool consistency. It is proposed to test both doses for the phase III program in chronic constipation.

The aim of this study is to demonstrate the effect of tegaserod on bowel habits in patients suffering from chronic idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria for entry into the study (Performed at screening):

* Male and females of at least 18 years of age (no upper limit).
* History of constipation for at least 12 months before screening. Constipation is defined as follows: less than three spontaneous bowel movements per week that result in a feeling of complete evacuation, and one or more of the following:

  * At least 25% of the stools are very hard and/or hard stools (Type 1 and/or 2 on the Bristol Stool Form scale)14,
  * Sensation of incomplete evacuation following at least 25% of the bowel movements
  * Straining on at least 25% of the defecations The above criteria are only applicable for spontaneous bowel movements, i.e. not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema. Patients who never have spontaneous bowel movements (that is, all bowel movements are preceded by laxatives) are considered constipated and eligible for the study.
* Patients who are able to communicate well with the investigator and to comply with the requirements for the entire study, including the withdrawal period.
* Patients who provide written informed consent before participating in the study after being given a full description of the study.

Exclusion Criteria for entry into the study (Performed at screening):

Patients meeting one or more of the following criteria should not be included in the study

* Use of herbs before 2 weeks of study
* Planned use of disallowed medication.
* With evidence of cathartic colon or a history of laxative abuse
* With a history of fecal impaction which necessitated surgical intervention
* Whose chronic constipation, according to the investigator's clinical judgment, is thought to be a result of: bowel surgery, gynecological surgery, neurologic disorders (e.g. aganglionosis, hypoganglionosis, autonomic neuropathy, Parkinson's disease, spinal cord injury or tumor, cerebrovascular accidents, multiple sclerosis), systemic sclerosis, myloidosis, scleroderma, myotonic dystrophy
* With a diagnosis of megarectum or colon, intestinal pseudo-obstruction, mechanical outlet obstruction, congenital anorectal malformation, rectocele, intestinal carcinoma, inlammatory bowel disease.
* An endoscopic/radiologic bowel evaluation (colonoscopic examination and/or a sigmoidoscopy + barium enema) is required in order to rule out cancer, inflammatory bowel disease or other structural disease. This evaluation must have been performed within the past 5 years. In addition, there should not be history or evidence of weight loss, anemia or rectal bleeding since the evaluation was performed.
* Existence of surgical or medical conditions which interfere with the absorption, distribution, metabolism and excretion of the study medication.
* With hypo or hyper thyroidism (clinically significant abnormal TSH level at screening)
* With clinical evidence (including physical exam, vital signs, ECG, laboratory tests) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematology, endocrine or metabolic disorders, neurologic disease, or of any disease that may interfere with the patient successfully completing the study . Patient with insulin-dependent diabetes are excluded from the study.
* With psychosis, schizophrenia, mania or major psychiatric illness needing pharmacological treatment. A well-compensated depression does not exclude a potential patient.
* With symptoms of a significant clinical illness in the two weeks preceding baseline.
* With other relevant intercurrent medical condition that may interfere with the objectives of the study.
* Women who are pregnant or breast-feeding.
* Fertile women who are not currently using or complying with a medically approved method of contraception such as, but not exclusively, one of the following:Oral birth control pills administered for at least 1 full monthly cycle prior to study medication administration, Progesterone implanted rods inserted for at least 1 month prior to study medication administration, Intra-uterine device (IUD), Medroxyprogesterone acetate administered for a minimum of 1 month prior to study medication administration and continued until 1 month following the last dose of study medication, Double barrier methods (such as condoms and spermicide), Abstinence, when in the opinion of the investigator, their occupation or life style gives sufficient evidence that abstinence will be maintained throughout the study and for 1 month thereafter. In the case of abstinence, it should be recorded in the source documents that the patient was appropriately counseled.

Fertile woman is defined as a woman who is not surgically sterile (i.e. hysterectomy, bilateral oophorectomy or bilateral tubal ligation), or is not post-menopausal (a post-menopausal patient is defined as a patient who has not menstruated for 12 months or more).

* With evidence or history of drug or alcohol abuse within the past 12 months.
* Who received another investigational drug within the 30 days prior to entry in the study.
* Who participated in a prior tegaserod study.

Exclusion criteria for randomization (Performed at Day 1):

Patients to be excluded from entry into the double-blind period of the study are those:

* Whose constipation, as defined in Inclusion Criteria No. 2, was not confirmed by the diary data of the baseline period (average of the last two weeks of baseline).
* With loose or watery stools (Type 6 or 7 stool form according to the Bristol stool form scale) occurring in more than 3 days during the baseline period.
* In whom exclusion criteria, listed for the baseline period, are identified prior to the start of the treatment period.
* Who did not comply with completing the daily diary assessments. To be randomized, a patient must have at least 11 days of complete daily diary data during the last 14 days of the baseline period.
* Who did not comply with completing the weekly diary assessments. To be randomized, a patient must have completed at least 1 complete weekly diary assessment during the last 14 days of the baseline period.
* Who deviated from the guidelines regarding prohibited medications (see section 3.4.4) more than two days (more than 3 days) during baseline.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
the response for the first 4 weeks of double-blind treatment period using the criterion based on the daily diary assessment | 4 Weeks

SECONDARY OUTCOMES:
Response rate throughout the 8 weeks of treatment | 8 Weeks
Evaluations of bowel habit | 12 Weeks
Patient' assessment of symptoms of constipation during the past week and Quality of life (QOL) assessment | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Annie OO Chan, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China